CLINICAL TRIAL: NCT03385434
Title: Evaluation of Endorings-2-assisted Colonoscopy: a New Accessory for Improvement of Adenoma Detection Rate?
Acronym: Endorings-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017-635-f-S
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colonic Adenoma; Colonic Polyp; Colonic Neoplasms; Colonoscopy
Keywords: Colonoscopy; adenoma detection rate; endorings-2; endorings; device-assisted colonoscopy
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endorings-assisted screening colonoscopy (Experimental): 146 patients with an indication for screening endoscopy will receive an Endorings-2-assisted colonoscopy.
  Interventions: Device: Endorings-2
- Standard screening colonoscopy (No Intervention): 146 patients with an indication for screening endoscopy will receive a standard colonoscopy.

INTERVENTIONS:
Device: Endorings-2 — 292 patients with an indication for screening colonoscopy will be included. 146 patients will receive a standard colonoscopy and 146 patients will receive an Endorings-2 assisted colonoscopy (1:1 standard colonoscopy vs Endorings-2-assisted colonoscopy).
  Other Names: Endorings-2 (EndoAid Ltd, Caesarea, Israel)
  Arms: Endorings-assisted screening colonoscopy

SUMMARY:
Screening colonoscopy for colorectal cancer is essential to diagnose and remove adenomas, precancerous stages of colorectal cancer. Unfortunately approximately 25 % of all adenomas are missed during the examination. Recently a new colonoscopy accessory, the Endorings-2 (EndoAid Ltd., Casearea, Israel), has been designed to improved the detection of adenomas during colonoscopy (adenoma detection rate).

Endorings-2 is a silicone-rubber device that is fitted on the colonoscope and is equipped with circular flexible silicon rings mechanically stretching the colonic folds during withdrawal.

This study aims to evaluate the efficacy of Endorings-2 to improve the adenoma detection rate in a prospective, blinded clinical trial. 292 patients with an indication for a screening colonoscopy shall be included (1:1 randomization in standard colonoscopy versus Endorings-2-assisted colonoscopy).

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for a screening colonoscopy.

Exclusion Criteria:

* Patients under 18 years, pregnancy
* Patients with prior colectomy or partial colectomy
* Patients with a history of colorectal cancer
* Patients with hereditary polyposis syndromes (FAP, HNPCC)
* Patients with a stricture of the colon
* Patients receiving anticoagulation prohibiting a colonoscopy
* inability to have a patient education
* bad conditions prohibiting a colonoscopy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the adenoma detection rate during screening colonoscopy | Intraoperative. Adenomas detected directly during the examination.
  The primary outcome of this study is the adenoma detection rate of the standard colonoscopy in comparison to the Endorings-assisted colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Unversity Clinic Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided